CLINICAL TRIAL: NCT01809041
Title: Comparison of Total Intravenous Anesthesia With Sevoflurane-based Balanced Anesthesia on Postoperative Cognitive Dysfunction in Elderly Patients for Major Elective Intra-abdominal Surgery
Brief Title: Comparison of Intravenous Anesthetics to Volatile Anesthetics on Postoperative Cognitive Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Huaqiao Hospital in Guangzhou, China (Other); First People's Hospital of Foshan (Other); Nanfang Hospital, Southern Medical University (Other); Guangdong Provincial People's Hospital, China (Unknown); Baxter (China) Investment Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Zhiyi Zuo, Visiting Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZZuo-POCD-1
Record Dates: First submitted 2013-03-06; First posted 2013-03-12 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Intra-abdominal and Intrapelvic Surgery
MeSH Terms: interventions — Sevoflurane; Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane & remifentanil (Experimental): sevoflurane at 0.5 to 1.5 minimum alveolar concentrations plus remifentanil (0.1 - 0.5 µg/kg/min) during the surgery.
  Interventions: Drug: Sevoflurane; Drug: remifentanil
- propofol & remifentanil (Active Comparator): propofol (50 - 150 µg/kg/min) and remifentanil (0.1 - 0.5 µg/kg/min)
  Interventions: Drug: propofol; Drug: remifentanil

INTERVENTIONS:
Drug: Sevoflurane
  Arms: Sevoflurane & remifentanil
Drug: propofol
  Arms: propofol & remifentanil
Drug: remifentanil

SUMMARY:
Post-operative cognitive dysfunction (POCD) is a fairly well-documented clinical phenomenon. Most patients will receive general anesthesia during surgery. Two groups of general anesthetics are used for this purpose. We hypothesize that the incidence of POCD is not different in patients received intravenous anesthetics only or sevoflurane (a volatile anesthetic-based general anesthesia) for their major intra-abdominal surgery.

DETAILED DESCRIPTION:
Patients who are 60 years old or older for laparoscopic abdominal surgery will be randomly assigned into two groups: 1) sevoflurane-based general anesthesia group, and 2) propofol-based general anesthesia group. Each group will need 221 patients to detect 1/3 of decrease or increase in the rate of POCD of one group compared with another group at about one week after surgery, assuming the overall rate of POCD at this time is about 40% at this time. Considering about 10% loss to follow-up, we will have 250 patients in each group. In addition, investigators will need 184 subjects in the control group. The data of these control subjects will be used to normalize the data of the two studied groups to diagnose POCD. The subjects in control groups will also be elderly but without the exposure to anesthesia and surgery.

ELIGIBILITY:
Inclusion Criteria:

1. major elective gastrointestinal, gynecological, prostate or bladder surgery patients who are ≥ 60 years old.
2. the surgery is laparoscopic surgery and is expected to last for ≥ 2 hours under general anesthesia and the patient will stay in hospital for at least 7 days after surgery.
3. lack of serious hearing and vision impairment and be able to read so that neurobehavioral tests can be performed.

Exclusion Criteria:

1. Patients are not expected to be alive for longer than 3 months.
2. Mini-mental State Examination (MMSE) [18] score ≤ 23.
3. history of dementia, psychiatric illness or any diseases of central nervous system.
4. current use of sedatives or antidepressant.
5. alcoholism and drug dependence.
6. patients previously included in this study (for patients who have second intra-abdominal surgery during the study period).
7. difficult to follow up or patients with poor compliance.
8. uncontrolled hypertension (> 180/100 mmHg)

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 684 (Estimated)
Dates: Start 2013-03; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with postoperative cognitive dysfunction (POCD) (POCD is a composite outcome measure) | At 7 days after the surgery
  Incidence of POCD in patients will be determined by a set of cognitive tests.

SECONDARY OUTCOMES:
Number of patients with postoperative cognitive dysfunction (POCD) (POCD is a composite outcome measure) | At 3 months after the surgery
  Incidence of POCD in patients will be determined by a set of cognitive tests.

OTHER OUTCOMES:
Time for bowel function return after surgery | up to 2 weeks after the surgery
  when bowel movement is returned.
Degree of increase of stress hormones | Up to 1 day after the surgery
  blood concentrations of stress hormones.
Length of hospital stay | Up to 3 months after the surgery
  duration of staying in the hospital
colorectal cancer progress | Up to one year after the surgery
  Migration, invasion and metastasis of the cancer
degree of systemic inflammation | Up to 7 days after surgery
  inflammatory cytokines in the blood
aging biochemical markers | Up to 7 days after surgery
  such as length of the telomere

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Background] Newman MF, Kirchner JL, Phillips-Bute B, Gaver V, Grocott H, Jones RH, Mark DB, Reves JG, Blumenthal JA; Neurological Outcome Research Group and the Cardiothoracic Anesthesiology Research Endeavors Investigators. Longitudinal assessment of neurocognitive function after coronary-artery bypass surgery. N Engl J Med. 2001 Feb 8;344(6):395-402. doi: 10.1056/NEJM200102083440601. PMID 11172175
- [Background] Steinmetz J, Christensen KB, Lund T, Lohse N, Rasmussen LS; ISPOCD Group. Long-term consequences of postoperative cognitive dysfunction. Anesthesiology. 2009 Mar;110(3):548-55. doi: 10.1097/ALN.0b013e318195b569. PMID 19225398
- [Background] Rasmussen LS, Johnson T, Kuipers HM, Kristensen D, Siersma VD, Vila P, Jolles J, Papaioannou A, Abildstrom H, Silverstein JH, Bonal JA, Raeder J, Nielsen IK, Korttila K, Munoz L, Dodds C, Hanning CD, Moller JT; ISPOCD2(International Study of Postoperative Cognitive Dysfunction) Investigators. Does anaesthesia cause postoperative cognitive dysfunction? A randomised study of regional versus general anaesthesia in 438 elderly patients. Acta Anaesthesiol Scand. 2003 Mar;47(3):260-6. doi: 10.1034/j.1399-6576.2003.00057.x. PMID 12648190
- [Background] Williams-Russo P, Sharrock NE, Mattis S, Szatrowski TP, Charlson ME. Cognitive effects after epidural vs general anesthesia in older adults. A randomized trial. JAMA. 1995 Jul 5;274(1):44-50. PMID 7791257